CLINICAL TRIAL: NCT00807976
Title: The Orthostatic Hypotension in the Diabetic Elderly Patients Trial (ODET)
Brief Title: Orthostatic Hypotension and Diabetes Mellitus
Acronym: ODET
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Kornelis J.J. van Hateren, Medical research foundation, The Netherlands
Other Study IDs: ODET1
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Orthostatic Hypotension; Diabetes Mellitus Type 2
Keywords: Diabetes mellitus; Elderly; Orthostatic hypotension
MeSH Terms: conditions — Hypotension, Orthostatic; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Type 2 diabetic patients aged 70 years and older.
- Control group: Patients aged 70 years and older, with no history of type 2 diabetes mellitus.

SUMMARY:
Rationale: Orthostatic hypotension increases with age and is associated with increased vascular and all-cause mortality. The prevalence of orthostatic hypotension is also increased in diabetic subjects. In order to prevent related adverse events and vascular mortality it is of great interest to examine the prevalence of orthostatic hypotension in elderly diabetic subjects.

Objective: To examine the prevalence of orthostatic hypotension and associated adverse events in type 2 diabetic elderly subjects.

Study design: Cross-sectional observational study.

Study population: Elderly type 2 diabetic subjects (70 years and older).

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* age (70 years and older)

Exclusion Criteria:

* Known autonomic dysfunction
* Neurodegenerative diseases
* Current malignancy
* Living in a nursing-home
* Irregular pulse

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Type 2 diabetic patients aged 70 years and older
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of orthostatic hypotension | 1-12 months (orthostatic blood pressure is assessed only once during the running time of the study)

SECONDARY OUTCOMES:
Adverse events, Score risk profile questionnaire, Heart rate, Gender, Body mass index, Medication, Smoking, History of cardiovascular disease, Family history of cardiovascular disease, Duration of diabetes mellitus, Glycosylated haemoglobin, Insulin use | 1-12 months (the outcome measures are assessed only once during the running time of the study)

CONTACTS AND LOCATIONS:
Overall Officials: Kornelis JJ van Hateren, MD, Principal Investigator — Diabetes centre, Isala Clinics
Locations (1):
- Diabetes centre, Isala Clinics, Zwolle, Netherlands